CLINICAL TRIAL: NCT04680819
Title: Evaluation of the Effect of Anatolian Propolis on Covid-19 in Healthcare Professionals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Principal Investigator, Ataturk University
Other Study IDs: AtaturkU2
Record Dates: First submitted 2020-12-19; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: covid-19; Anatolian Propolis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compared with given anatolian propolis group and do not use anatolian propolis group: According to the spectrophotometic analysis report of this anatolian group, there should be a minimum phenolic 106.0 mg gae per ml and 73.1 mg ke flavonoid content in each ml and a total content of 253.9 mg te / ml.
  Interventions: Dietary Supplement: Anatolian Propolis

INTERVENTIONS:
Dietary Supplement: Anatolian Propolis — Health workers who agree to participate in the study will be accepted as the study group, and healthcare professionals who do not agree to participate in the study will be considered as the control group. The study group will be asked to take 20 drops of Propolis drop form twice a day in the morning / evening, and the control group will not receive any treatment and both groups will be followed. In this process, patients diagnosed with COVID-19 will be determined. PCR test positivity taken from the throat for the diagnosis of COVID-19 will be accepted. The research will cover a period of 1 month. At the end of 1 month, patients diagnosed with COVID-19 in the study and control groups will be compared. Thus, the protective properties of Anatolian propolis will be determined.

SUMMARY:
There is no prophylaxis for people at high risk of developing COVID-19. It is one of the first clinical studies aiming to investigate the effect of Anatolian Propolis against COVID-19. This study will test whether Anatolian propolis can be used to prevent the development of COVID-19 in people at risk of COVID-19. If Anatolian Propolis has been shown to reduce the risk of developing COVID-19 in people at high risk of infection, this could help reduce the morbidity and mortality of the COVID-19 outbreak.

This study will be done in 2 centers. These centers are planned as Atatürk University Medical Faculty Emergency Medicine Clinic and Rize Recep Tayyip Erdoğan University Emergency Medicine Clinic. This work will be done entirely on a voluntary basis. The research subject will be explained to the healthcare professionals (doctor, nurse, medical secretary) working in both emergency medicine clinics and voluntary participation forms will be signed by the healthcare professionals who agree to participate in the study. Health workers who agree to participate in the study will be accepted as the study group, and healthcare professionals who do not agree to participate in the study will be accepted as the control group. The study group will be asked to take 20 drops of Propolis drop form twice a day in the morning / evening and the control group will not receive any treatment and both groups will be followed. In this process, patients diagnosed with COVID-19 will be determined.The study will cover a period of 1 month and at the end of 1 month, patients diagnosed with COVID-19 in the study and control groups will be compared. Thus, the protective properties of Anatolian propolis will be determined.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome Coronavirus - 2 (SARS-CoV-2) caused by Covid-19 epidemics have been implicated in 330,000 more than cases in Turkey and 40 health workers at a rate close to 5% by thousand cases affected by this epidemic and There is a serious increase in risk for people every day.

There is currently no established post-exposure prophylaxis for people at high risk of developing COVID-19. Propolis, a natural resin produced by bees and of plant origin, has anti-inflammatory, immunomodulatory, anti-oxidant properties, and various aspects of the SARS-CoV-2 infection mechanism are potential targets for propolis compounds. This work; It is a randomized study aiming to evaluate the effect of Anatolian propolis extract against the effects of the new coronavirus threatening human health. In this clinical study, the product containing Anatolian propolis will be used to evaluate its effectiveness. According to the spectrophotometic analysis report of this product, there should be a minimum phenolic 106.0 mg gae per ml and 73.1 mg ke flavonoid content in each ml and a total content of 253.9 mg te / ml.

There is no prophylaxis for people at high risk of developing COVID-19. It is one of the first clinical studies aiming to investigate the effect of Anatolian Propolis against COVID-19. This study will test whether Anatolian propolis can be used to prevent the development of COVID-19 in people at risk of COVID-19. If Anatolian Propolis has been shown to reduce the risk of developing COVID-19 in people at high risk of infection, this could help reduce the morbidity and mortality of the COVID-19 outbreak.

This study will be done in 2 centers. These centers are planned as Atatürk University Medical Faculty Emergency Medicine Clinic and Rize Recep Tayyip Erdoğan University Emergency Medicine Clinic. This work will be done entirely on a voluntary basis. The research subject will be explained to the healthcare professionals (doctor, nurse, medical secretary) working in both emergency medicine clinics and voluntary participation forms will be signed by the healthcare professionals who agree to participate in the study. Health workers who agree to participate in the study will be accepted as the study group, and healthcare professionals who do not agree to participate in the study will be accepted as the control group. The study group will be asked to take 20 drops of Propolis drop form twice a day in the morning / evening and the control group will not receive any treatment and both groups will be followed. In this process, patients diagnosed with COVID-19 will be determined.

For the diagnosis of COVID-19, PCR test positivity taken from the throat will be accepted. The study will cover a period of 1 month and at the end of 1 month, patients diagnosed with COVID-19 in the study and control groups will be compared. Thus, the protective properties of Anatolian propolis will be determined.

The data obtained will be analyzed with the SPSS.20 program. Data will be given as percentages and numbers. Shapiro-Wilk and Kolmogorov-Smirnov tests will be used to evaluate whether the data are suitable for normal distribution. Independent samples t-test will be used to compare data normally distributed between two independent groups, and the Mann-Whitney U test will be used if the data are not normally distributed. Categorical variables will be compared using Chi-square and Fisher tests. A value of p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Not having had COVID-19 (diagnosed by PCR)
* Symptom that may be associated with COVID-19 for the past 14 days (fever, fatigue, loss of taste and smell)
* No additional chronic disease (such as chronic heart lung)
* Healthcare workers (doctor, nurse, medical secretary)
* Working in an emergency medicine clinic
* Being a volunteer

Exclusion Criteria:

* Not being willing to participate in research
* Patients younger than 18 years old,
* Pregnant patients
* Immunosuppressive patients
* Patients receiving chemotherapy for any reason
* Being appointed to another clinic from the emergency medicine clinic within a 1-month period planned as a working period
* Propolis allergy or history of hypersensitivity to any of its ingredients.
* Volunteers taking a break from drug use during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy emergency room workers who volunteer to participate in the research
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-25 (Estimated); Primary Completion 2021-01-25 (Estimated); Study Completion 2021-01-25 (Estimated)

PRIMARY OUTCOMES:
Covid-19 positive | 1 month
  For the diagnosis of COVID-19, the positivity of the PCR test taken from the throat will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Ataturk University Osman, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: Yes
will be shared as soon as appropriate.
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: completion of the article